CLINICAL TRIAL: NCT00737269
Title: A Prospective, Multi-center, Observational Registry Involving Patients Hospitalized With Complicated Skin and Soft Tissue Infections (cSSTI) for IV Antibiotic Therapy
Brief Title: A Complicated Skin and Soft-tissue Infection Patient Registry
Status: Completed | Type: Observational
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015043; CEFTOSSK4001 (Other: Ortho-McNeil Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Staphylococcal Skin Infections; Diabetic Foot Infections; Surgical Wound Infection; Abscess; Cellulitis
Keywords: Complicated Skin and Soft-Tissue Infection; Skin Infection; Skin Infection Registry; cSSTI Registry
MeSH Terms: conditions — Staphylococcal Skin Infections; Surgical Wound Infection; Abscess; Cellulitis; Soft Tissue Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this registry is to better understand (1) complicated skin and soft-tissue infections requiring hospitalization, and (2) clinical and economic outcomes in hospitalized patients receiving intravenous antibiotic therapy.

DETAILED DESCRIPTION:
A prospective, multi-center, observational study involving 1200 patients hospitalized for the treatment of cSSTIs. The study will be conducted at approximately 50 hospitals in the US. Patients who consent to participate in the registry will be enrolled in the registry within 24 hours of initial IV antibiotic therapy for treatment of one or more cSSTI types. Sites will treat patients according to their usual clinical practice. The objective of this registry is to characterize cSSTIs with respect to patient characteristics and describe patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of complicated skin and soft-tissue infection
* Patients who require IV antibiotic therapy as a primary treatment regimen
* Patients who are deemed to be cognitive and able to provide written informed consent and follow-up information.

Exclusion Criteria:

* Patients with a diagnosis at the index infection site of necrotizing soft tissue infection, burn, gangrene, decubitus ulcer, animal or human bites, known or suspected osteomyelitis, or mediastinitis
* Patients for whom amputation or a complete resection of the infection site is a planned component of treatment
* Patients who are pregnant
* Patients simultaneously participating in any interventional clinical trial
* Patients with any other known or suspected condition that may jeopardize adherence to registry protocol requirements
* Patients who are employees of the investigator or study hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complicated skin and soft tissue infections (specifically, diabetic foot infections, surgical site infections, deep soft tissue abscess, cellulitis)
Sampling Method: Non-Probability Sample
Enrollment: 1081 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC